CLINICAL TRIAL: NCT00626093
Title: Effect of Cardiac Resynchronization Therapy (CRT) on the Defibrillation Threshold (DFT) Estimates
Brief Title: 'Effect of CRT on Defibrillation Threshold Estimates' Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD 388
Record Dates: First submitted 2008-02-07; First posted 2008-02-29 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Sudden Cardiac Death
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac Resynchronization Therapy - Defibrillator (CRT-D) (Other): Patients in the study who received a Cardiac Resynchronization Therapy - Defibrillator (CRT-D) are indicated for it. It's a single arm study in which patients underwent defibrillation threshold (DFT) testing at implant and 6 months.
  Interventions: Device: Cardiac Resynchronization Therapy - Defibrillator (CRT-D)

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy - Defibrillator (CRT-D) — * Patients in the study who receive Cardiac Resynchronization Therapy - Defibrillator (CRT-D) are indicated for Cardiac Resynchronization Therapy (CRT).
  * Patient undergoes Defibrillation threshold (DFT) testing at implant and at 6 months. Defibrillation threshold (DFT) testing will include 3 ventricular fibrillation (VF) inductions.
  Other Names: Epic HF,Atlas+ HF,Epic II HF,Atlas II HF,Promote CRT-D

SUMMARY:
The purpose of this prospective study is to evaluate the effect of cardiac resynchronization therapy (CRT) on the defibrillation threshold (DFT) estimates in cardiac resynchronization therapy defibrillators (CRT-D) patients. The hypothesis of the study is that defibrillation threshold (DFT) will decrease with 6 months of cardiac resynchronization therapy (CRT).

DETAILED DESCRIPTION:
Cardiac Resynchronization Therapy (CRT) has emerged as a promising therapeutic addition in patients with drug refractory heart failure (HF). Along with providing relief of symptoms of HF, cardiac resynchronization therapy defibrillators (CRT-D) are used for the prevention of sudden cardiac death (SCD). Although there are concerns that the defibrillation threshold (DFT) estimates are elevated in the heart failure (HF) patient population due to lower LV ejection fraction (EF) and left ventricular (LV) dysfunction, there is paucity of data available to evaluate this theory.

Recently, two different studies in a retrospective manner evaluated the energy requirements in patients receiving cardiac resynchronization therapy defibrillators (CRT-D). Burke et al analyzed DFTs in 50 patients each implanted with a cardiac resynchronization therapy defibrillators (CRT-D) device and an implantable cardioverter defibrillator (ICD). Although the ejection fraction (EF) in cardiac resynchronization therapy defibrillators (CRT- D) group was lower than the implantable cardioverter defibrillator (ICD) group, the mean defibrillation thresholds (DFTs) between the two groups were not significantly different (10.2 ± 6.1 J for the cardiac resynchronization therapy (CRT) group vs. 9.5 ± 5.0 J for the control group)14. In the ASSURE study, Doshi et al. showed that patients receiving cardiac resynchronization therapy defibrillators (CRT-D) devices do not have higher energy requirements when compared to patients receiving modern single or dual chamber implantable cardioverter defibrillators (ICDs). Although, there was a trend toward higher energy requirements found among patients with higher degrees of heart failure.

Major cardiac resynchronization therapy (CRT) trials have showed that cardiac resynchronization therapy (CRT) therapy has positive effects on ejection fraction (EF) and the heart failure (HF) condition of the patient over time. But, there is no study that has evaluated the defibrillation thresholds (DFTs) in the heart failure (HF) patients over time of receiving cardiac resynchronization therapy (CRT). This information will help the clinicians decide if they need to perform more invasive procedures during device implant to lower DFTs in patients who do not meet the defibrillation safety margin or they should just wait over time for the CRT to reduce the defibrillation threshold (DFT). Also, there is no published data about the stability of defibrillation thresholds (DFTs) in heart failure (HF) patients over time. The results from this study will also help to clarify whether it is safe to never test the defibrillation thresholds (DFTs) post-implant in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets standard indications for a Cardiac Resynchronization Therapy - Defibrillator (CRT-D).
* Patient will be implanted with an FDA approved St Jude Medical (SJM) Cardiac Resynchronization Therapy - Defibrillator (CRT-D) and compatible defibrillation lead system.
* Patient is able to tolerate defibrillation threshold (DFT) testing.
* Patient is geographically stable and willing to comply with the required follow-up schedule.
* Patient has a life expectancy of greater than 6 months from the time of implant.
* Patient has stable heart failure (HF) medications at least one month prior to enrollment.

Exclusion Criteria:

* Inability to successfully implant an intravascular lead Cardiac Resynchronization Therapy - Defibrillator (CRT-D) device. (i.e. exclude epicardial leads).
* Patient is getting his Cardiac Resynchronization Therapy - Defibrillator (CRT-D) device replaced.
* Inability to successfully obtain the defibrillation threshold (DFT) at implant.
* Currently participating in a clinical trial that includes an active treatment arm or another data collection registry.
* Recent (within 24 hours) administration of Nesiritide™.
* Patient is on amiodarone (other antiarrhythmic agents known to affect defibrillation thresholds - DFTs) at the time of enrollment.
* Patient is pregnant.
* Patient is less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Hedayati, MD, Principal Investigator — Glendale Heart Institute; Michael Gold, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Pacific Heart Institute, Santa Monica, California
  - Penrose Hospital, Colorado Springs, Colorado

REFERENCES:
- [Result] Gold MR, Hedayati A, Alaeddini J, Payne JP, Bailin S, Sturdivant JJ, Pradhan S, Oza AL. Temporal stability of defibrillation thresholds with cardiac resynchronization therapy. Heart Rhythm. 2011 Jul;8(7):1008-13. doi: 10.1016/j.hrthm.2011.02.006. Epub 2011 Feb 9. PMID 21315841

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardiac Resynchronization Therapy - Defibrillators (CRT-D): All patients enrolled were indicated for a CRT-D.
Period: Overall Study
Arm/Group | Cardiac Resynchronization Therapy - Defibrillators (CRT-D)
Started | 77
Completed | 54
Not Completed | 23
Not completed — Lost to Follow-up | 5
Not completed — Death | 1
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 1
Not completed — One of the required devices not implante | 6

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 54
Region of Enrollment [Number; unit: participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Defibrillation Threshold Difference Obtained in Volts (V) Between Implant and 6 Months
Description: All patients underwent defibrillation threshold testing at cardiac resynchronization therapy-defibrillator (CRT-D) implant and then at 6 months. The outcome measure is the difference in DFT (defibrillation threshold) in volts between implant and 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | CRT-D
Number analyzed (Participants) | 77
Volts | 5.6 (110.5)

2. Secondary Outcome: Defibrillation Threshold Difference Obtained in Joules (J)
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Joules
Arm/Group | CRT-D
Number analyzed (Participants) | 77
Joules | 0.3 (5)

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 1/77
Other Adverse Events (participants affected / at risk) | 4/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=77)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=77)
Phrenic Nerve Stimulation (Cardiac disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No